CLINICAL TRIAL: NCT03132636
Title: A Phase 2 Study of REGN2810, a Fully Human Monoclonal Antibody to Programmed Death-1, in Patients With Advanced Basal Cell Carcinoma Who Experienced Progression of Disease on Hedgehog Pathway Inhibitor Therapy, or Were Intolerant of Prior Hedgehog Pathway Inhibitor Therapy
Brief Title: PD-1 in Patients With Advanced Basal Cell Carcinoma Who Experienced Progression of Disease on Hedgehog Pathway Inhibitor Therapy, or Were Intolerant of Prior Hedgehog Pathway Inhibitor Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R2810-ONC-1620; 2016-003122-16 (EudraCT Number)
Record Dates: First submitted 2017-04-24; First posted 2017-04-28 (Actual); Results first posted 2022-07-26 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Carcinoma, Basal Cell
MeSH Terms: conditions — Carcinoma, Basal Cell | interventions — cemiplimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group 1- metastatic BCC (Experimental): Administration of cemiplimab in accordance with protocol dosing regimen
  Interventions: Drug: cemiplimab
- Group 2 - unresectable locally advanced BCC (Experimental): Administration of cemiplimab in accordance with protocol dosing regimen
  Interventions: Drug: cemiplimab

INTERVENTIONS:
Drug: cemiplimab — Regimen as per protocol
  Other Names: REGN2810; Libtayo

SUMMARY:
The primary objective is to estimate the objective response rate (ORR) for metastatic Basal Cell Carcinoma (BCC) (group 1) and for unresectable locally advanced BCC (group 2) when treated with cemiplimab as a monotherapy

ELIGIBILITY:
Key Inclusion Criteria:

* Confirmed diagnosis of invasive BCC
* Progression of disease on hedgehog inhibitor (HHI) therapy or intolerance of prior HHI therapy
* At least 1 measurable lesion
* ≥18 years of age
* Hepatic function, renal function, bone marrow function in defined lab-value-ranges
* Anticipated life expectancy >12 weeks
* Consent to provide archived tumor biopsy material (all patients)
* Group 2: consent to undergo research biopsies
* Group 2: must not be a candidate for radiation therapy or surgery
* Comply with study procedures and site visits
* Sign Subject Information Sheet and Informed Consent Form

Key Exclusion Criteria:

* Ongoing or recent significant autoimmune disease
* Prior treatment with specific pathway-blockers (PD-1/PD-L1)
* Prior treatment with immune-modulating agents within 28 days before cemiplimab
* Untreated brain metastasis that may be considered active
* Immunosuppressive corticosteroid doses (>10mg prednisone) within 28 days prior to treatment with cemiplimab
* Active infections requiring therapy, including HIV, hepatitis
* Pneumonitis within the last 5 years
* Cancer treatment other than radiation therapy, including investigational or standard of care, within 30 days prior to treatment with cemiplimab
* Documented allergic reactions or similar to antibody treatments
* Concurrent malignancies other than BCC, other than those with negligible risk of metastases or death
* Any acute or chronic psychiatric problems
* Having received a solid organ transplantation
* Inability to undergo contrast radiological assessments
* Breastfeeding, pregnant, women of childbearing potential not using contraception

Note: Other protocol-defined inclusion/exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2017-06-29 (Actual); Primary Completion 2021-05-20 (Actual); Study Completion 2023-04-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (71):
- United States (23):
  - The University of Arizona Cancer Centre at Dignity Health, Phoenix, Arizona
  - Mayo Clinic Arizona - Mayo Clinic Hospital, Phoenix, Arizona
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Stanford Medicine Outpatient Center - Stanford Dermatology Clinic-Stanford University School of Medicine, Redwood City, California
  - UCSF Helen Dillion Family Cancer Care Center, San Francisco, California
  - University of Colorado Hospital, Anschutz Outpatient Pavilion, Denver, Colorado
  - Mount Sinai Comprehensive Cancer Center, Miami, Florida
  - H Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Northwestern Medical Faculty Foundation, Chicago, Illinois
  - Norton Cancer Institute, Louisville, Kentucky
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute (DFCI), Boston, Massachusetts
  - Washington University School of Medicine, St Louis, Missouri
  - Atlantic Health System / Morristown Medical Center, Morristown, New Jersey
  - Overlook Medical Center, Summit, New Jersey
  - New York University School Of Medicine, Kaplan Comprehensive Cancer Center, New York, New York
  - Mount Sinai Hospital, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - James Cancer Hospital and Solove Research Institute, Columbus, Ohio
  - Penn State Hershey Medical Center, Hershey, Pennsylvania
  - Clinical Research Center of the Carolinas, Charleston, South Carolina
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
- Austria (2):
  - LKH - Universitaetsklinikum Graz, Graz, Styria
  - Medizinische Universitaet Innsbruck, Universitaetsklinik fuer Dermatologie, Venerologie und Allergologie, Innsbruck
- Belgium (2):
  - Cliniques Universitaires Saint-Luc, Brussels
  - Universitaire Ziekenhuizen Leuven - Campus Gasthuisberg, Leuven
- Canada (4):
  - Cross Cancer Institute, Edmonton, Alberta
  - Odette Cancer Center-Sunnybrook Health Sciences Centre, Toronto, Ontario
  - University Health Network, Toronto, Ontario
  - London Regional Cancer Program, London Hsc, Toronto, Ontario
- France (12):
  - CHU de Dijon - Hopital du Bocage, Dijon, Cedex
  - Hopital Saint Louis, Paris, Europe
  - Centre Hospitalier Lyon-Sud -Hospices Civils de Lyon Groupement Hospitalier Sud, Pierre-Bénite, Paris
  - Centre Hospitalier Universitaire de Bordeaux - Groupe Hospitalier Saint-André - Hôpital Saint-André, Bordeaux
  - Hopital Ambroise Pare, Boulogne-Billancourt
  - Centre Hospitalier Universitaire de Grenoble, La Tronche
  - Hopital Huriez - CHRU de Lille, Lille
  - Centre Leon-Berard (CLB), Lyon
  - CHU Hotel Dieu, Nantes
  - Centre Hospitalier Universitaire de Rouen-Hopital Charles Nicolle, Rouen
  - Institut Claudius Regaud, Toulouse
  - Institut Gustave Roussy, Villejuif
- Germany (12):
  - University Hospital Frankfurt, Frankfurt, Hessen/Germany
  - Hauttumorcentrum der Charite (HTCC)-Charite Universitatsmedizin Berlin, Berlin
  - Elbekliniken Buxtehude, Buxtehude
  - University Hospital Dresden, Dresden
  - Universitaetsklinik Essen, Essen
  - SRH Wald-Kliniken Gera GmbH, Gera
  - Hannover Medical School, Hanover
  - NCT Dermatoonkologie, Heidelberg
  - University of Kiel, Kiel
  - Universitaetsmedizin der Johannes Gutenberg-Universitaet Mainz, Mainz
  - Klinik Fur Dermatologie Und Allergollogie, Quedlinburg
  - University Hospital Tubingen, Tübingen
- Greece (4):
  - National and Kapodistrian University of Athens - School of Health Sciences - Faculty of Medicine, Athens
  - National and Kapodistrian University of Athens - School of Health Sciences, Athens
  - Andreas Sygros Hosptial-University of Athen, Athens
  - University General Hospital of Ioannina - Dermatology and Venereology Department, Ioannina
- Italy (7):
  - Policlinico S.Orsola-Malpighi U.O. Dermatologia - University of Bologna, Bologna, Bo
  - Azienda Ospedaliera Spedali Civili di Brescia-Universita degli Studi Di Brescia, Brescia, Province Of Brescia
  - U.O.Dermatologia Azienda Sanitaria Firenze Universita' Firenze, Florence
  - University L'Aquila, L’Aquila
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan
  - U.O.S.C Di Oncologia Medica E Terapie Innovative, Napoli
  - Catholic University of the S.Heart, Roma
- Spain (4):
  - Catalan Institute of Oncology Badalona, Badalona
  - Hospital Clinic I Provincialde Barcelona, Barcelona
  - Hospital Universitario de Torrejon, Madrid
  - Hospital Universitario Virgen Macarena, Seville
- University Hospital Zurich Usz, Zurich, Switzerland

REFERENCES:
- [Derived] Stratigos AJ, Chen CI, Ivanescu C, Lewis KD, Peris K, Bechter O, Harnett J, Mastey V, Reaney M, Daskalopoulou C, LaFontaine PR, Konidaris G, Bury D, Yoo SY, Mohan K, Coates E, Bowler T, Fury MG, Sekulic A. Quality of life in cemiplimab-treated patients with locally advanced basal cell carcinoma in a Phase II clinical trial. Future Oncol. 2024;20(30):2249-2258. doi: 10.1080/14796694.2024.2358670. Epub 2024 Jul 29. PMID 39073799
- [Derived] Lewis KD, Peris K, Sekulic A, Stratigos AJ, Dunn L, Eroglu Z, Chang ALS, Migden MR, Yoo SY, Mohan K, Coates E, Okoye E, Bowler T, Baurain JF, Bechter O, Hauschild A, Butler MO, Hernandez-Aya L, Licitra L, Neves RI, Ruiz ES, Seebach F, Lowy I, Goncalves P, Fury MG. Final analysis of phase II results with cemiplimab in metastatic basal cell carcinoma after hedgehog pathway inhibitors. Ann Oncol. 2024 Feb;35(2):221-228. doi: 10.1016/j.annonc.2023.10.123. Epub 2023 Dec 9. PMID 38072158
- [Derived] Stratigos AJ, Sekulic A, Peris K, Bechter O, Prey S, Lewis KD, Basset-Seguin N, Chang ALS, Dalle S, Fernandez Orland A, Licitra L, Robert C, Ulrich C, Hauschild A, Migden MR, Dummer R, Yoo SY, Okoye E, Bassukas I, Loquai C, De Giorgi V, Eroglu Z, Gutzmer R, Ulrich J, Puig S, Inocencio TJ, Chen CI, LaFontaine PR, Seebach F, Lowy I, Fury MG. Phase 2 open-label, multicenter, single-arm study of cemiplimab in patients with locally advanced basal cell carcinoma after hedgehog inhibitor therapy: Extended follow-up. J Am Acad Dermatol. 2024 Feb;90(2):414-418. doi: 10.1016/j.jaad.2023.08.111. Epub 2023 Oct 14. No abstract available. PMID 37839734
- [Derived] Stratigos AJ, Sekulic A, Peris K, Bechter O, Prey S, Kaatz M, Lewis KD, Basset-Seguin N, Chang ALS, Dalle S, Orland AF, Licitra L, Robert C, Ulrich C, Hauschild A, Migden MR, Dummer R, Li S, Yoo SY, Mohan K, Coates E, Jankovic V, Fiaschi N, Okoye E, Bassukas ID, Loquai C, De Giorgi V, Eroglu Z, Gutzmer R, Ulrich J, Puig S, Seebach F, Thurston G, Weinreich DM, Yancopoulos GD, Lowy I, Bowler T, Fury MG. Cemiplimab in locally advanced basal cell carcinoma after hedgehog inhibitor therapy: an open-label, multi-centre, single-arm, phase 2 trial. Lancet Oncol. 2021 Jun;22(6):848-857. doi: 10.1016/S1470-2045(21)00126-1. Epub 2021 May 14. PMID 34000246
- [Derived] Li R, Lee G, Huang M, El-Sherief A. Rare basal cell metastasis of a basal-squamous skin collision tumour to the lung and axillary lymph node. BMJ Case Rep. 2019 Oct 3;12(10):e231487. doi: 10.1136/bcr-2019-231487. PMID 31585957
- See also: A Plain Language Summary is available on TrialSummaries.com — https://www.trialsummaries.com/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 138 of the 170 screened participants, were enrolled & treated. Eligible participants were enrolled into 2 groups. Group 1: participants with metastatic Basal Cell Carcinoma (mBCC). Group 2: participants with unresectable locally advanced BCC (laBCC) who experienced progression of disease on Hedgehog inhibitor (HHI) therapy, or response no better than stable disease for at least 9 months or were intolerant of prior HHI therapy.
Groups:
- Group 1: Metastatic BCC (mBCC): Participants with metastatic BCC received IV infusion of cemiplimab at a dose of 350 mg Q3W for up to 93 weeks of treatment cycles (cycles 1-5 [each cycle of 9 weeks] followed by cycles 6-9 [each cycle of 12 weeks]) or until PD, unacceptable toxicity, withdrawal of consent, or CR.
- Group 2: Unresectable Locally Advanced BCC (laBCC): Participants with unresectable laBCC received IV infusion of cemiplimab at a dose of 350 mg Q3W for up to 93 weeks of treatment cycles (cycles 1-5 [each cycle of 9 weeks] followed by cycles 6-9 [each cycle of 12 weeks]) or until PD, unacceptable toxicity, withdrawal of consent, or confirmed CR.
Period: Overall Study
Arm/Group | Group 1: Metastatic BCC (mBCC) | Group 2: Unresectable Locally Advanced BCC (laBCC)
Started | 54 | 84
Completed Treatment | 11 | 28
Completed (Completed Study) | 6 | 19
Not Completed | 48 | 65
Not completed — Adverse Event | 1 | 2
Not completed — Death | 4 | 7
Not completed — Lost to Follow-up | 3 | 2
Not completed — Non compliance with protocol by participant | 1 | 1
Not completed — Subject decision | 1 | 9
Not completed — Sponsor decision | 0 | 1
Not completed — Physician Decision | 1 | 0
Not completed — Progressive disease | 33 | 36
Not completed — Withdrawal of consent | 2 | 5
Not completed — Did not re-consent | 1 | 0
Not completed — Lost insurance coverage | 1 | 0
Not completed — Related to radiological outcomes | 0 | 1
Not completed — Unable to come to site for continued visits | 0 | 1

BASELINE CHARACTERISTICS:
Population: The full analysis set (FAS) included all enrolled participants for each group who passed screening and were deemed to be eligible for this study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: Metastatic BCC (mBCC) | Group 2: Unresectable Locally Advanced BCC (laBCC) | Total
Number analyzed (Participants) | 54 | 84 | 138
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.8 (11.09) | 69.1 (12.84) | 67.0 (12.42)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 28 | 44
  Male | 38 | 56 | 94
Race/Ethnicity, Customized [Number; unit: Participants]
  Race : White | 47 | 57 | 104
  Race : Not Reported | 1 | 0 | 1
  Race : Missing | 6 | 27 | 33
Race/Ethnicity, Customized [Number; unit: Participants]
  Ethnicity : Not Hispanic or Latino | 46 | 56 | 102
  Ethnicity : Hispanic or Latino | 2 | 1 | 3
  Ethnicity : Missing | 6 | 27 | 33

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR) as Assessed by Independent Central Review (ICR)
Description: ORR was defined as percentage of participants with best overall response of complete response (CR) or partial response (PR) according to RECIST v1.1 assessed as per ICR assessment. CR: Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to less than (<) 10 millimeter (mm) (< 1 centimeter [cm]). PR: At least a 30 percent (%) decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters. ORR was determined by Clopper-Pearson method.
Time Frame: Up to 1422 days (approximately 46 months)
Population: Full analysis set (FAS) (included all enrolled participants for each group who passed screening and were deemed to be eligible for this study)
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Group 1: Metastatic BCC (mBCC) | Group 2: Unresectable Locally Advanced BCC (laBCC)
Number analyzed (Participants) | 54 | 84
Percentage of Participants | 22.2 [12.0 to 35.6] | 32.1 [22.4 to 43.2]

2. Secondary Outcome: Objective Response Rate (ORR) Per Investigator Assessment
Description: ORR was defined as percentage of participants with best overall response of complete response (CR) or partial response (PR) according to RECIST v1.1 per Investigator assessment. CR: Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to less than (<) 10 millimeter (mm) (< 1 centimeter [cm]). PR: At least a 30 percent (%) decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters. ORR was determined by Clopper-Pearson method.
Time Frame: Up to 1422 days (approximately 46 months)
Population: The FAS included all enrolled participants for each group who passed screening and were deemed to be eligible for this study.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Group 1: Metastatic BCC (mBCC) | Group 2: Unresectable Locally Advanced BCC (laBCC)
Number analyzed (Participants) | 54 | 84
Percentage of Participants | 25.9 [15.0 to 39.7] | 36.9 [26.6 to 48.1]

3. Secondary Outcome: Duration of Response (DOR) as Assessed by ICR
Description: DOR per ICR was determined for participants with best overall response of CR or PR. DOR was measured from the time measurement criteria are first met for CR/PR (whichever was first recorded) until the first date of recurrent or progressive disease (PD) (photographic or radiographic), or death due to any cause. CR: Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm (<1 cm). PR: At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters. PD: At least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). DOR was determined by Kaplan-Meier estimate.
Time Frame: Up to 48 months
Population: The FAS included all enrolled participants for each group who passed screening and were deemed to be eligible for this study. Here, "Overall number of participants analyzed" signifies those participants with confirmed CR or PR.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Group 1: Metastatic BCC (mBCC) | Group 2: Unresectable Locally Advanced BCC (laBCC)
Number analyzed (Participants) | 12 | 27
Months | NA [9.8 to NA] — Because 50.0% of participants were censored and there was a greater than 50% chance of surviving at follow-up, the median survival and upper bounds of the 95% confidence interval could not be estimated. | NA [15.5 to NA] — Because 70.4% of participants were censored and there was a greater than 50% chance of surviving at follow-up, the median survival and upper bounds of the 95% confidence interval could not be estimated.

4. Secondary Outcome: Duration of Response (DOR) Per Investigator Assessment
Description: DOR per investigator assessment was determined for participants with best overall response of CR or PR. DOR was measured from the time measurement criteria are first met for CR/PR (whichever was first recorded) until the first date of recurrent or progressive disease (PD) (photographic or radiographic), or death due to any cause. CR: Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm (<1 cm). PR: At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters. PD: At least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). DOR was determined by Kaplan-Meier estimate.
Time Frame: Up to 48 months
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Group 1: Metastatic BCC (mBCC) | Group 2: Unresectable Locally Advanced BCC (laBCC)
Number analyzed (Participants) | 14 | 31
Months | NA [9.8 to NA] — Data could not be estimated due to higher number (64.3%) of censored participants | 19.6 [16.7 to NA] — Data could not be estimated due to higher number (54.8%) of censored participants

5. Secondary Outcome: Complete Response (CR) Rate as Assessed by ICR
Description: CR rate was determined by the percentage of participants with best overall response of CR. CR: Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm (<1 cm). CR rate 95% confidence interval determined by Clopper-Pearson exact confidence interval.
Time Frame: Up to 48 months
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Group 1: Metastatic BCC (mBCC) | Group 2: Unresectable Locally Advanced BCC (laBCC)
Number analyzed (Participants) | 54 | 84
Percentage of Participants | 3.7 [0.5 to 12.7] | 8.3 [3.4 to 16.4]

6. Secondary Outcome: Complete Response (CR) Rate Per Investigator Assessment
Description: as for outcome 5
Time Frame: Up to 48 months
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Group 1: Metastatic BCC (mBCC) | Group 2: Unresectable Locally Advanced BCC (laBCC)
Number analyzed (Participants) | 54 | 84
Percentage of Participants | 3.7 [0.5 to 12.7] | 8.3 [3.4 to 16.4]

7. Secondary Outcome: Progression Free Survival (PFS) as Assessed by ICR
Description: PFS was defined as the time from start of treatment until the first date of recurrent or PD (photographic or radiographic), or death due to any cause, whichever occurred first, was determined by IRC. PD: At least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). PFS was determined by Kaplan-Meier estimate.
Time Frame: Up to 60 months
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Group 1: Metastatic BCC (mBCC) | Group 2: Unresectable Locally Advanced BCC (laBCC)
Number analyzed (Participants) | 54 | 84
Months | 10.1 [4.2 to 15.9] | 16.5 [8.6 to 21.8]

8. Secondary Outcome: Progression Free Survival (PFS) Per Investigator Assessment
Description: as for outcome 7
Time Frame: Up to 60 months
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Group 1: Metastatic BCC (mBCC) | Group 2: Unresectable Locally Advanced BCC (laBCC)
Number analyzed (Participants) | 54 | 84
Months | 6.6 [4.2 to 8.3] | 18.1 [10.4 to 21.3]

9. Secondary Outcome: Overall Survival (OS)
Description: OS was measured as time from the start of treatment until death due to any cause. Participants who did not die were censored at the last date that participant was documented to be alive. OS was calculated based on Kaplan-Meier estimate.
Time Frame: Up to 60 months
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Group 1: Metastatic BCC (mBCC) | Group 2: Unresectable Locally Advanced BCC (laBCC)
Number analyzed (Participants) | 54 | 84
Months | 49.9 [28.4 to NA] — Because 59.3% of participants were censored and there was a greater than 50% chance of surviving at follow-up, the upper bound of the 95% confidence interval could not be estimated. | NA [NA to NA] — Because 75.0% of participants were censored and there was a greater than 50% chance of surviving at follow-up, the median overall survival and lower and upper bounds of the 95% confidence interval could not be estimated.

10. Secondary Outcome: Change From Baseline of Patient-reported Outcomes in European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30)
Description: The EORTC QLQ-C30 is a 30-item questionnaire used to assess the overall QoL in cancer participants. It consists of 15 domains: 1 Global Health Status (GHS)/QoL scale, 5 functional scales (Physical, role, cognitive, emotional, social), 9 symptom scales/items (Fatigue, nausea and vomiting, pain, dyspnea, sleep disturbance, appetite loss, constipation, diarrhea, financial impact). Most items are scored 1 ("not at all") to 4 ("very much") except for the items contributing to the GHS/QoL, which are scored 1 ("very poor") to 7 ("excellent"). A linear transformation was applied to the raw scores so that all transformed scores lie between 0 to 100. For the GHS/QoL and 5 functional scales a higher score indicates higher ("better") quality of life/functioning and a positive change from baseline indicates improvement. For the symptom scales/items, a higher score indicates a higher ("worse") level of symptoms/problems, and a negative change from baseline indicates improvement.
Time Frame: Baseline (Day 1 of Cycle 1); Day 1 of Cycles 2 to 9 (Cycles 1-5 [Each cycle of 9 weeks], Cycles 6 to 9 [Each cycle of 12 weeks])
Population: The FAS included all enrolled participants for each group who passed screening and were deemed to be eligible for this study. "Number analyzed" signifies those participants who were evaluable at specific time points.
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Group 1: Metastatic BCC (mBCC) | Group 2: Unresectable Locally Advanced BCC (laBCC)
Number analyzed (Participants) | 54 | 84
Score on a Scale
  Physical Functioning: Change at Cycle 2 Day 1: number analyzed (Participants) | 43 | 75
  Physical Functioning: Change at Cycle 2 Day 1 | -4.88 (14.274) | -1.55 (12.101)
  Physical Functioning: Change at Cycle 3 Day 1: number analyzed (Participants) | 29 | 65
  Physical Functioning: Change at Cycle 3 Day 1 | -1.78 (13.481) | -0.56 (15.947)
  Physical Functioning: Change at Cycle 4 Day 1: number analyzed (Participants) | 26 | 55
  Physical Functioning: Change at Cycle 4 Day 1 | -6.60 (12.828) | -3.79 (17.814)
  Physical Functioning: Change at Cycle 5 Day 1: number analyzed (Participants) | 20 | 50
  Physical Functioning: Change at Cycle 5 Day 1 | 1.08 (10.033) | -2.86 (17.063)
  Physical Functioning: Change at Cycle 6 Day 1: number analyzed (Participants) | 19 | 40
  Physical Functioning: Change at Cycle 6 Day 1 | -1.67 (9.734) | 0.33 (12.073)
  Physical Functioning: Change at Cycle 7 Day 1: number analyzed (Participants) | 13 | 33
  Physical Functioning: Change at Cycle 7 Day 1 | -0.38 (11.142) | -0.20 (15.410)
  Physical Functioning: Change at Cycle 8 Day 1: number analyzed (Participants) | 10 | 33
  Physical Functioning: Change at Cycle 8 Day 1 | -1.33 (12.090) | -3.03 (13.549)
  Physical Functioning: Change at Cycle 9 Day 1: number analyzed (Participants) | 11 | 29
  Physical Functioning: Change at Cycle 9 Day 1 | -2.27 (8.765) | -5.06 (20.444)
  Role Functioning: Change at Cycle 2 Day 1 | -2.71 (27.442) | -3.11 (20.264)
  Role Functioning: Change at Cycle 3 Day 1: number analyzed (Participants) | 29 | 65
  Role Functioning: Change at Cycle 3 Day 1 | 5.17 (27.854) | -4.87 (25.297)
  Role Functioning: Change at Cycle 4 Day 1: number analyzed (Participants) | 26 | 55
  Role Functioning: Change at Cycle 4 Day 1 | -3.21 (25.394) | -6.06 (26.326)
  Role Functioning: Change at Cycle 5 Day 1: number analyzed (Participants) | 20 | 50
  Role Functioning: Change at Cycle 5 Day 1 | 5.00 (22.361) | -5.33 (26.393)
  Role Functioning: Change at Cycle 6 Day 1: number analyzed (Participants) | 19 | 40
  Role Functioning: Change at Cycle 6 Day 1 | 6.14 (21.667) | -3.33 (16.963)
  Role Functioning: Change at Cycle 7 Day 1: number analyzed (Participants) | 13 | 33
  Role Functioning: Change at Cycle 7 Day 1 | 12.82 (24.677) | -7.07 (16.682)
  Role Functioning: Change at Cycle 8 Day 1: number analyzed (Participants) | 10 | 33
  Role Functioning: Change at Cycle 8 Day 1 | 15.00 (25.398) | -4.04 (19.557)
  Role Functioning: Change at Cycle 9 Day 1: number analyzed (Participants) | 11 | 29
  Role Functioning: Change at Cycle 9 Day 1 | 9.09 (22.808) | -9.77 (30.052)
  Emotional Functioning: Change at Cycle 2 Day 1: number analyzed (Participants) | 54 | 74
  Emotional Functioning: Change at Cycle 2 Day 1 | 3.17 (19.638) | 1.95 (20.483)
  Emotional Functioning: Change at Cycle 3 Day 1: number analyzed (Participants) | 29 | 64
  Emotional Functioning: Change at Cycle 3 Day 1 | 1.15 (18.730) | 1.56 (18.538)
  Emotional Functioning: Change at Cycle 4 Day 1: number analyzed (Participants) | 26 | 54
  Emotional Functioning: Change at Cycle 4 Day 1 | 3.53 (22.007) | 1.39 (21.277)
  Emotional Functioning: Change at Cycle 5 Day 1: number analyzed (Participants) | 20 | 49
  Emotional Functioning: Change at Cycle 5 Day 1 | 5.83 (24.046) | -4.59 (19.622)
  Emotional Functioning: Change at Cycle 6 Day 1: number analyzed (Participants) | 19 | 40
  Emotional Functioning: Change at Cycle 6 Day 1 | 7.02 (20.650) | 1.04 (19.809)
  Emotional Functioning: Change at Cycle 7 Day 1: number analyzed (Participants) | 13 | 33
  Emotional Functioning: Change at Cycle 7 Day 1 | 3.85 (18.199) | -4.63 (19.576)
  Emotional Functioning: Change at Cycle 8 Day 1: number analyzed (Participants) | 11 | 33
  Emotional Functioning: Change at Cycle 8 Day 1 | 16.67 (25.000) | 3.11 (19.810)
  Emotional Functioning: Change at Cycle 9 Day 1: number analyzed (Participants) | 11 | 29
  Emotional Functioning: Change at Cycle 9 Day 1 | 5.30 (17.189) | 2.11 (17.246)
  Cognitive Functioning: Change at Cycle 2 Day 1: number analyzed (Participants) | 54 | 74
  Cognitive Functioning: Change at Cycle 2 Day 1 | 0.78 (13.586) | -2.48 (26.985)
  Cognitive Functioning: Change at Cycle 3 Day 1: number analyzed (Participants) | 29 | 64
  Cognitive Functioning: Change at Cycle 3 Day 1 | -1.72 (16.871) | -4.17 (23.382)
  Cognitive Functioning: Change at Cycle 4 Day 1: number analyzed (Participants) | 26 | 54
  Cognitive Functioning: Change at Cycle 4 Day 1 | -0.64 (15.261) | -4.94 (21.385)
  Cognitive Functioning: Change at Cycle 5 Day 1: number analyzed (Participants) | 20 | 49
  Cognitive Functioning: Change at Cycle 5 Day 1 | -4.17 (14.178) | -6.46 (25.188)
  Cognitive Functioning: Change at Cycle 6 Day 1: number analyzed (Participants) | 19 | 40
  Cognitive Functioning: Change at Cycle 6 Day 1 | -0.88 (12.998) | -1.25 (19.017)
  Cognitive Functioning: Change at Cycle 7 Day 1: number analyzed (Participants) | 13 | 33
  Cognitive Functioning: Change at Cycle 7 Day 1 | -2.56 (11.479) | -5.56 (18.942)
  Cognitive Functioning: Change at Cycle 8 Day 1: number analyzed (Participants) | 11 | 33
  Cognitive Functioning: Change at Cycle 8 Day 1 | -6.06 (11.237) | 1.52 (17.362)
  Cognitive Functioning: Change at Cycle 9 Day 1: number analyzed (Participants) | 11 | 29
  Cognitive Functioning: Change at Cycle 9 Day 1 | -10.61 (25.025) | -2.30 (23.873)
  Social Functioning: Change at Cycle 2 Day 1: number analyzed (Participants) | 54 | 74
  Social Functioning: Change at Cycle 2 Day 1 | 0.39 (19.412) | 4.50 (21.422)
  Social Functioning: Change at Cycle 3 Day 1: number analyzed (Participants) | 29 | 64
  Social Functioning: Change at Cycle 3 Day 1 | 3.45 (16.891) | 0.78 (21.088)
  Social Functioning: Change at Cycle 4 Day 1: number analyzed (Participants) | 26 | 54
  Social Functioning: Change at Cycle 4 Day 1 | 3.85 (24.179) | 1.85 (23.272)
  Social Functioning: Change at Cycle 5 Day 1: number analyzed (Participants) | 20 | 49
  Social Functioning: Change at Cycle 5 Day 1 | 3.33 (22.685) | 0.34 (23.445)
  Social Functioning: Change at Cycle 6 Day 1: number analyzed (Participants) | 19 | 40
  Social Functioning: Change at Cycle 6 Day 1 | 10.53 (16.860) | 0.00 (24.749)
  Social Functioning: Change at Cycle 7 Day 1: number analyzed (Participants) | 13 | 33
  Social Functioning: Change at Cycle 7 Day 1 | 12.82 (22.724) | 0.00 (18.162)
  Social Functioning: Change at Cycle 8 Day 1: number analyzed (Participants) | 11 | 33
  Social Functioning: Change at Cycle 8 Day 1 | 10.61 (15.407) | 2.02 (23.848)
  Social Functioning: Change at Cycle 9 Day 1: number analyzed (Participants) | 11 | 29
  Social Functioning: Change at Cycle 9 Day 1 | 9.09 (13.670) | -2.30 (27.359)
  Fatigue: Change at Cycle 2 Day 1 | 5.17 (22.919) | 6.44 (24.542)
  Fatigue: Change at Cycle 3 Day 1: number analyzed (Participants) | 29 | 65
  Fatigue: Change at Cycle 3 Day 1 | 1.92 (18.322) | 6.58 (24.901)
  Fatigue: Change at Cycle 4 Day 1: number analyzed (Participants) | 26 | 55
  Fatigue: Change at Cycle 4 Day 1 | -2.56 (21.154) | 7.58 (25.912)
  Fatigue: Change at Cycle 5 Day 1: number analyzed (Participants) | 20 | 50
  Fatigue: Change at Cycle 5 Day 1 | -5.56 (24.048) | 9.67 (23.404)
  Fatigue: Change at Cycle 6 Day 1: number analyzed (Participants) | 19 | 40
  Fatigue: Change at Cycle 6 Day 1 | -5.85 (19.376) | 7.78 (17.649)
  Fatigue: Change at Cycle 7 Day 1: number analyzed (Participants) | 13 | 33
  Fatigue: Change at Cycle 7 Day 1 | -1.71 (19.692) | 14.14 (20.838)
  Fatigue: Change at Cycle 8 Day 1: number analyzed (Participants) | 10 | 33
  Fatigue: Change at Cycle 8 Day 1 | -7.78 (24.595) | 9.09 (19.534)
  Fatigue: Change at Cycle 9 Day 1: number analyzed (Participants) | 11 | 29
  Fatigue: Change at Cycle 9 Day 1 | -1.01 (16.067) | 12.64 (20.080)
  Nausea/Vomiting: Change at Cycle 2 Day 1 | -0.78 (8.095) | 0.22 (12.703)
  Nausea/Vomiting: Change at Cycle 3 Day 1: number analyzed (Participants) | 29 | 65
  Nausea/Vomiting: Change at Cycle 3 Day 1 | 0.00 (13.363) | -1.79 (12.884)
  Nausea/Vomiting: Change at Cycle 4 Day 1: number analyzed (Participants) | 26 | 55
  Nausea/Vomiting: Change at Cycle 4 Day 1 | 0.00 (16.330) | 0.30 (13.414)
  Nausea/Vomiting: Change at Cycle 5 Day 1: number analyzed (Participants) | 20 | 50
  Nausea/Vomiting: Change at Cycle 5 Day 1 | 0.83 (10.080) | 1.00 (13.640)
  Nausea/Vomiting: Change at Cycle 6 Day 1: number analyzed (Participants) | 19 | 40
  Nausea/Vomiting: Change at Cycle 6 Day 1 | -0.88 (3.824) | 1.67 (13.503)
  Nausea/Vomiting: Change at Cycle 7 Day 1: number analyzed (Participants) | 13 | 33
  Nausea/Vomiting: Change at Cycle 7 Day 1 | -1.28 (14.372) | 3.03 (13.472)
  Nausea/Vomiting: Change at Cycle 8 Day 1: number analyzed (Participants) | 10 | 33
  Nausea/Vomiting: Change at Cycle 8 Day 1 | 0.00 (0.000) | 0.51 (12.832)
  Nausea/Vomiting: Change at Cycle 9 Day 1: number analyzed (Participants) | 11 | 29
  Nausea/Vomiting: Change at Cycle 9 Day 1 | 0.00 (0.000) | -2.30 (13.890)
  Pain: Change at Cycle 2 Day 1 | -2.33 (30.338) | -0.22 (26.351)
  Pain: Change at Cycle 3 Day 1: number analyzed (Participants) | 29 | 65
  Pain: Change at Cycle 3 Day 1 | -9.77 (22.056) | -1.54 (30.151)
  Pain: Change at Cycle 4 Day 1: number analyzed (Participants) | 26 | 55
  Pain: Change at Cycle 4 Day 1 | 0.00 (29.439) | -4.85 (25.795)
  Pain: Change at Cycle 5 Day 1: number analyzed (Participants) | 20 | 50
  Pain: Change at Cycle 5 Day 1 | -4.17 (25.291) | -4.00 (25.098)
  Pain: Change at Cycle 6 Day 1: number analyzed (Participants) | 19 | 40
  Pain: Change at Cycle 6 Day 1 | -14.04 (29.535) | -2.92 (24.427)
  Pain: Change at Cycle 7 Day 1: number analyzed (Participants) | 13 | 33
  Pain: Change at Cycle 7 Day 1 | -21.79 (29.174) | -4.04 (24.661)
  Pain: Change at Cycle 8 Day 1: number analyzed (Participants) | 11 | 33
  Pain: Change at Cycle 8 Day 1 | -13.64 (25.624) | -7.58 (25.716)
  Pain: Change at Cycle 9 Day 1: number analyzed (Participants) | 11 | 29
  Pain: Change at Cycle 9 Day 1 | -19.70 (27.707) | -5.17 (24.030)
  Dyspnoea: Change at Cycle 2 Day 1: number analyzed (Participants) | 42 | 84
  Dyspnoea: Change at Cycle 2 Day 1 | 2.38 (17.097) | 1.33 (24.162)
  Dyspnoea: Change at Cycle 3 Day 1: number analyzed (Participants) | 28 | 65
  Dyspnoea: Change at Cycle 3 Day 1 | 3.57 (16.578) | -0.51 (23.930)
  Dyspnoea: Change at Cycle 4 Day 1: number analyzed (Participants) | 25 | 55
  Dyspnoea: Change at Cycle 4 Day 1 | 0.00 (16.667) | 2.42 (24.724)
  Dyspnoea: Change at Cycle 5 Day 1: number analyzed (Participants) | 19 | 49
  Dyspnoea: Change at Cycle 5 Day 1 | 3.51 (21.928) | 0.00 (28.054)
  Dyspnoea: Change at Cycle 6 Day 1: number analyzed (Participants) | 18 | 40
  Dyspnoea: Change at Cycle 6 Day 1 | 1.85 (13.873) | -1.67 (19.900)
  Dyspnoea: Change at Cycle 7 Day 1: number analyzed (Participants) | 12 | 33
  Dyspnoea: Change at Cycle 7 Day 1 | 2.78 (30.011) | 2.02 (21.952)
  Dyspnoea: Change at Cycle 8 Day 1: number analyzed (Participants) | 10 | 33
  Dyspnoea: Change at Cycle 8 Day 1 | 16.67 (36.004) | 2.02 (21.952)
  Dyspnoea: Change at Cycle 9 Day 1: number analyzed (Participants) | 10 | 29
  Dyspnoea: Change at Cycle 9 Day 1 | 6.67 (26.294) | 2.30 (17.663)
  Insomnia: Change at Cycle 2 Day 1 | -2.33 (26.622) | 0.44 (24.195)
  Insomnia: Change at Cycle 3 Day 1: number analyzed (Participants) | 29 | 65
  Insomnia: Change at Cycle 3 Day 1 | -6.90 (24.200) | -0.51 (26.016)
  Insomnia: Change at Cycle 4 Day 1: number analyzed (Participants) | 26 | 55
  Insomnia: Change at Cycle 4 Day 1 | -10.26 (29.468) | -1.82 (19.687)
  Insomnia: Change at Cycle 5 Day 1: number analyzed (Participants) | 20 | 50
  Insomnia: Change at Cycle 5 Day 1 | -15.00 (31.484) | 1.33 (30.087)
  Insomnia: Change at Cycle 6 Day 1: number analyzed (Participants) | 19 | 40
  Insomnia: Change at Cycle 6 Day 1 | -17.54 (32.142) | -4.17 (24.093)
  Insomnia: Change at Cycle 7 Day 1: number analyzed (Participants) | 13 | 33
  Insomnia: Change at Cycle 7 Day 1 | -7.69 (41.172) | 1.01 (28.241)
  Insomnia: Change at Cycle 8 Day 1: number analyzed (Participants) | 10 | 33
  Insomnia: Change at Cycle 8 Day 1 | -13.33 (54.885) | 3.03 (25.500)
  Insomnia: Change at Cycle 9 Day 1: number analyzed (Participants) | 11 | 29
  Insomnia: Change at Cycle 9 Day 1 | -6.06 (38.925) | 5.75 (25.306)
  Appetite loss: Change at Cycle 2 Day 1: number analyzed (Participants) | 54 | 74
  Appetite loss: Change at Cycle 2 Day 1 | 4.65 (26.807) | -2.25 (27.215)
  Appetite loss: Change at Cycle 3 Day 1: number analyzed (Participants) | 29 | 62
  Appetite loss: Change at Cycle 3 Day 1 | -2.30 (15.252) | -4.30 (22.163)
  Appetite loss: Change at Cycle 4 Day 1: number analyzed (Participants) | 26 | 54
  Appetite loss: Change at Cycle 4 Day 1 | -1.28 (30.523) | -3.09 (26.117)
  Appetite loss: Change at Cycle 5 Day 1: number analyzed (Participants) | 20 | 49
  Appetite loss: Change at Cycle 5 Day 1 | 3.33 (21.357) | -1.36 (30.398)
  Appetite loss: Change at Cycle 6 Day 1: number analyzed (Participants) | 19 | 39
  Appetite loss: Change at Cycle 6 Day 1 | -1.75 (17.476) | -2.56 (29.004)
  Appetite loss: Change at Cycle 7 Day 1: number analyzed (Participants) | 13 | 33
  Appetite loss: Change at Cycle 7 Day 1 | -5.13 (12.518) | -1.01 (30.601)
  Appetite loss: Change at Cycle 8 Day 1: number analyzed (Participants) | 10 | 32
  Appetite loss: Change at Cycle 8 Day 1 | -3.33 (10.541) | -2.08 (31.609)
  Appetite loss: Change at Cycle 9 Day 1: number analyzed (Participants) | 11 | 28
  Appetite loss: Change at Cycle 9 Day 1 | -3.03 (17.979) | 1.19 (30.741)
  Constipation: Change at Cycle 2 Day 1: number analyzed (Participants) | 54 | 74
  Constipation: Change at Cycle 2 Day 1 | 1.55 (19.181) | 2.25 (21.603)
  Constipation: Change at Cycle 3 Day 1: number analyzed (Participants) | 29 | 63
  Constipation: Change at Cycle 3 Day 1 | 0.00 (21.822) | 1.06 (20.712)
  Constipation: Change at Cycle 4 Day 1: number analyzed (Participants) | 26 | 54
  Constipation: Change at Cycle 4 Day 1 | -2.56 (18.674) | 1.23 (21.440)
  Constipation: Change at Cycle 5 Day 1: number analyzed (Participants) | 20 | 49
  Constipation: Change at Cycle 5 Day 1 | 5.00 (16.312) | -0.68 (22.037)
  Constipation: Change at Cycle 6 Day 1: number analyzed (Participants) | 19 | 40
  Constipation: Change at Cycle 6 Day 1 | 0.00 (15.713) | -1.67 (18.413)
  Constipation: Change at Cycle 7 Day 1: number analyzed (Participants) | 13 | 33
  Constipation: Change at Cycle 7 Day 1 | 5.13 (18.490) | 4.04 (13.838)
  Constipation: Change at Cycle 8 Day 1: number analyzed (Participants) | 10 | 33
  Constipation: Change at Cycle 8 Day 1 | 13.33 (23.307) | -2.02 (16.540)
  Constipation: Change at Cycle 9 Day 1: number analyzed (Participants) | 11 | 29
  Constipation: Change at Cycle 9 Day 1 | 0.00 (14.907) | 1.15 (22.683)
  Diarhoea: Change at Cycle 2 Day 1: number analyzed (Participants) | 54 | 74
  Diarhoea: Change at Cycle 2 Day 1 | 3.88 (14.924) | 0.45 (24.360)
  Diarhoea: Change at Cycle 3 Day 1: number analyzed (Participants) | 29 | 64
  Diarhoea: Change at Cycle 3 Day 1 | 1.15 (14.037) | -1.04 (20.547)
  Diarhoea: Change at Cycle 4 Day 1: number analyzed (Participants) | 26 | 54
  Diarhoea: Change at Cycle 4 Day 1 | 3.85 (23.715) | -1.85 (19.870)
  Diarhoea: Change at Cycle 5 Day 1: number analyzed (Participants) | 20 | 49
  Diarhoea: Change at Cycle 5 Day 1 | 6.67 (20.520) | -0.68 (23.064)
  Diarhoea: Change at Cycle 6 Day 1: number analyzed (Participants) | 19 | 40
  Diarhoea: Change at Cycle 6 Day 1 | 3.51 (18.904) | -1.67 (18.413)
  Diarhoea: Change at Cycle 7 Day 1: number analyzed (Participants) | 13 | 33
  Diarhoea: Change at Cycle 7 Day 1 | 0.00 (13.608) | 1.01 (19.516)
  Diarhoea: Change at Cycle 8 Day 1: number analyzed (Participants) | 11 | 33
  Diarhoea: Change at Cycle 8 Day 1 | 0.00 (14.907) | -1.01 (19.516)
  Diarhoea: Change at Cycle 9 Day 1: number analyzed (Participants) | 11 | 29
  Diarhoea: Change at Cycle 9 Day 1 | 0.00 (14.907) | -2.30 (21.696)
  Financial Problems: Change at Cycle 2 Day 1: number analyzed (Participants) | 54 | 74
  Financial Problems: Change at Cycle 2 Day 1 | -3.10 (17.539) | -3.15 (25.385)
  Financial Problems: Change at Cycle 3 Day 1: number analyzed (Participants) | 28 | 63
  Financial Problems: Change at Cycle 3 Day 1 | 0.00 (18.144) | -4.23 (24.313)
  Financial Problems: Change at Cycle 4 Day 1: number analyzed (Participants) | 26 | 54
  Financial Problems: Change at Cycle 4 Day 1 | -5.13 (22.494) | -4.94 (23.710)
  Financial Problems: Change at Cycle 5 Day 1: number analyzed (Participants) | 20 | 49
  Financial Problems: Change at Cycle 5 Day 1 | 0.00 (18.732) | -6.80 (22.546)
  Financial Problems: Change at Cycle 6 Day 1: number analyzed (Participants) | 19 | 40
  Financial Problems: Change at Cycle 6 Day 1 | -1.75 (23.501) | -5.83 (27.099)
  Financial Problems: Change at Cycle 7 Day 1: number analyzed (Participants) | 13 | 33
  Financial Problems: Change at Cycle 7 Day 1 | -2.56 (21.350) | 1.01 (19.516)
  Financial Problems: Change at Cycle 8 Day 1: number analyzed (Participants) | 11 | 33
  Financial Problems: Change at Cycle 8 Day 1 | -3.03 (17.979) | 1.01 (19.516)
  Financial Problems: Change at Cycle 9 Day 1: number analyzed (Participants) | 11 | 29
  Financial Problems: Change at Cycle 9 Day 1 | -6.06 (20.101) | -2.30 (23.454)
  Global health status/QoL: Change at Cycle 2 Day 1: number analyzed (Participants) | 54 | 72
  Global health status/QoL: Change at Cycle 2 Day 1 | -3.68 (21.845) | 2.55 (15.298)
  Global health status/QoL: Change at Cycle 3 Day 1: number analyzed (Participants) | 29 | 62
  Global health status/QoL: Change at Cycle 3 Day 1 | 3.74 (14.362) | -2.55 (19.823)
  Global health status/QoL: Change at Cycle 4 Day 1: number analyzed (Participants) | 26 | 51
  Global health status/QoL: Change at Cycle 4 Day 1 | -2.24 (14.636) | -0.49 (18.136)
  Global health status/QoL: Change at Cycle 5 Day 1: number analyzed (Participants) | 20 | 48
  Global health status/QoL: Change at Cycle 5 Day 1 | 7.50 (14.023) | -1.91 (21.210)
  Global health status/QoL: Change at Cycle 6 Day 1: number analyzed (Participants) | 19 | 38
  Global health status/QoL: Change at Cycle 6 Day 1 | 10.96 (11.802) | 4.17 (19.447)
  Global health status/QoL: Change at Cycle 7 Day 1: number analyzed (Participants) | 13 | 32
  Global health status/QoL: Change at Cycle 7 Day 1 | 16.03 (22.428) | -3.13 (19.715)
  Global health status/QoL: Change at Cycle 8 Day 1: number analyzed (Participants) | 11 | 31
  Global health status/QoL: Change at Cycle 8 Day 1 | 9.09 (13.670) | 2.15 (21.727)
  Global health status/QoL: Change at Cycle 9 Day 1: number analyzed (Participants) | 11 | 28
  Global health status/QoL: Change at Cycle 9 Day 1 | 8.33 (20.412) | -7.14 (28.211)

11. Secondary Outcome: Change From Baseline of Patient-reported Outcomes in Skindex-16 Questionnaire
Description: Skindex-16 questionnaire contains 16 questions related to quality of life in cancer participants. It consisted of a short 16-item assessment completed by the participant, with each item rated on a 7-point Likert scale (0=never bothered to 6=always bothered). Each raw score is multiplied by 16.667 to transform all responses to a linear scale from 0 (no effect) to 100 (effect experienced all the time). Responses to the Skindex-16 are categorized into 3 subscales: symptom, emotional & functional; their respective scores are expressed in a linear scale from 0 to 100. Symptoms scale score was an average of items 1 to 4 expressed in a linear scale from 0 to 100, Emotions scale score was an average of items 5 to 11 expressed in a linear scale from 0 to 100 and Functioning scale score was an average of items 12 to 16 expressed in a linear scale from 0 to 100. A negative change from baseline indicates an improvement in the participants condition compared to the baseline.
Time Frame: as for outcome 10
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Group 1: Metastatic BCC (mBCC) | Group 2: Unresectable Locally Advanced BCC (laBCC)
Number analyzed (Participants) | 54 | 84
Score on a Scale
  Emotions: Change at Cycle 2 Day 1: number analyzed (Participants) | 42 | 69
  Emotions: Change at Cycle 2 Day 1 | -6.90 (24.422) | -8.93 (27.767)
  Emotions: Change at Cycle 3 Day 1: number analyzed (Participants) | 26 | 63
  Emotions: Change at Cycle 3 Day 1 | -7.92 (18.033) | -8.60 (25.641)
  Emotions: Change at Cycle 4 Day 1: number analyzed (Participants) | 22 | 51
  Emotions: Change at Cycle 4 Day 1 | -3.97 (17.175) | -11.45 (24.215)
  Emotions: Change at Cycle 5 Day 1: number analyzed (Participants) | 17 | 46
  Emotions: Change at Cycle 5 Day 1 | -0.14 (12.835) | -10.25 (24.646)
  Emotions: Change at Cycle 6 Day 1: number analyzed (Participants) | 16 | 35
  Emotions: Change at Cycle 6 Day 1 | -9.08 (22.824) | -19.73 (27.304)
  Emotions: Change at Cycle 7 Day 1: number analyzed (Participants) | 12 | 30
  Emotions: Change at Cycle 7 Day 1 | 6.55 (17.053) | -13.65 (27.132)
  Emotions: Change at Cycle 8 Day 1: number analyzed (Participants) | 10 | 30
  Emotions: Change at Cycle 8 Day 1 | -0.71 (8.478) | -13.97 (25.001)
  Emotions: Change at Cycle 9 Day 1: number analyzed (Participants) | 11 | 28
  Emotions: Change at Cycle 9 Day 1 | 5.70 (14.711) | -15.08 (31.843)
  Symptoms: Change at Cycle 2 Day 1 | 0.99 (18.788) | -1.31 (21.607)
  Symptoms: Change at Cycle 3 Day 1: number analyzed (Participants) | 26 | 64
  Symptoms: Change at Cycle 3 Day 1 | 3.85 (16.580) | -0.26 (24.158)
  Symptoms: Change at Cycle 4 Day 1: number analyzed (Participants) | 22 | 52
  Symptoms: Change at Cycle 4 Day 1 | 5.30 (18.464) | -6.62 (23.917)
  Symptoms: Change at Cycle 5 Day 1: number analyzed (Participants) | 17 | 47
  Symptoms: Change at Cycle 5 Day 1 | -0.98 (15.205) | -4.11 (18.062)
  Symptoms: Change at Cycle 6 Day 1: number analyzed (Participants) | 16 | 36
  Symptoms: Change at Cycle 6 Day 1 | -1.56 (16.307) | -1.85 (21.419)
  Symptoms: Change at Cycle 7 Day 1: number analyzed (Participants) | 12 | 30
  Symptoms: Change at Cycle 7 Day 1 | 4.17 (23.233) | 0.69 (24.518)
  Symptoms: Change at Cycle 8 Day 1: number analyzed (Participants) | 10 | 31
  Symptoms: Change at Cycle 8 Day 1 | 5.00 (17.213) | -2.96 (24.395)
  Symptoms: Change at Cycle 9 Day 1: number analyzed (Participants) | 11 | 28
  Symptoms: Change at Cycle 9 Day 1 | 8.33 (21.246) | -3.42 (24.455)
  Functioning: Change at Cycle 2 Day 1 | -3.49 (19.183) | -4.98 (23.650)
  Functioning: Change at Cycle 3 Day 1: number analyzed (Participants) | 26 | 63
  Functioning: Change at Cycle 3 Day 1 | -5.00 (18.166) | -4.76 (20.203)
  Functioning: Change at Cycle 4 Day 1: number analyzed (Participants) | 22 | 51
  Functioning: Change at Cycle 4 Day 1 | -8.18 (24.119) | -5.82 (23.275)
  Functioning: Change at Cycle 5 Day 1: number analyzed (Participants) | 17 | 47
  Functioning: Change at Cycle 5 Day 1 | -7.06 (20.746) | -3.76 (16.369)
  Functioning: Change at Cycle 6 Day 1: number analyzed (Participants) | 16 | 35
  Functioning: Change at Cycle 6 Day 1 | -12.08 (27.022) | -11.14 (18.113)
  Functioning: Change at Cycle 7 Day 1: number analyzed (Participants) | 12 | 30
  Functioning: Change at Cycle 7 Day 1 | -3.89 (19.583) | -6.00 (15.767)
  Functioning: Change at Cycle 8 Day 1: number analyzed (Participants) | 10 | 30
  Functioning: Change at Cycle 8 Day 1 | -7.33 (23.402) | -7.00 (17.926)
  Functioning: Change at Cycle 9 Day 1: number analyzed (Participants) | 11 | 28
  Functioning: Change at Cycle 9 Day 1 | -9.39 (21.072) | -5.60 (20.965)

12. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Serious TEAEs
Description: An adverse event (AE) was defined as any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. TEAEs are defined as AEs that developed or worsened during the on-treatment period and treatment-related AEs that occur during post-treatment period. A serious adverse event (SAE) was defined as any untoward medical occurrence that resulted in any of the following outcomes: death, life-threatening, required initial or prolonged in-patient hospitalization, persistent or significant disability/incapacity, congenital anomaly/birth defect, or considered as medically important event. Any TEAE included participants with both serious and non-serious TEAEs.
Time Frame: Up to 1422 days (approximately 46 months)
Population: The safety analysis set (SAF) included all enrolled participants who received any study drug for each group.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Metastatic BCC (mBCC) | Group 2: Unresectable Locally Advanced BCC (laBCC)
Number analyzed (Participants) | 54 | 84
Participants
  Participants with any TEAEs | 51 | 83
  Participants with any Serious TEAEs | 16 | 31

13. Secondary Outcome: Serum Concentration at Pre-infusion (Ctrough)
Description: Ctrough of cemiplimab reported.
Time Frame: At pre-infusion on Cycle 1 Day 22 and Cycle 3 Day 1 (Each cycle of 9 weeks)
Population: The PK analysis set included all participants who received any cemiplimab and had at least one non-missing post-baseline measurement of cemiplimab concentration in serum. "Number analyzed" signifies those participants who were evaluable at specific time points.
Measure: Mean (Standard Deviation); unit: Milligram per Liter (mg/L)
Arm/Group | Group 1: Metastatic BCC (mBCC) | Group 2: Unresectable Locally Advanced BCC (laBCC)
Number analyzed (Participants) | 54 | 84
Milligram per Liter (mg/L)
  Cycle 1 Day 22: number analyzed (Participants) | 50 | 78
  Cycle 1 Day 22 | 28.3 (18.4) | 29.8 (12.0)
  Cycle 3 Day 1: number analyzed (Participants) | 32 | 66
  Cycle 3 Day 1 | 60.6 (28.2) | 68.6 (32.8)

14. Secondary Outcome: Serum Concentration at End of Infusion (Cmax)
Description: Cmax of cemiplimab was reported.
Time Frame: At end-of-infusion (within 10 minutes after the end of infusion) on Cycle 1 Day 1 and Cycle 3 Day 1 (Each cycle of 9 weeks)
Population: The pharmacokinetics (PK) analysis set included all participants who received any cemiplimab and had at least one non-missing post-baseline measurement of cemiplimab concentration in serum. "Number analyzed" signifies those participants who were evaluable at specific time points.
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Group 1: Metastatic BCC (mBCC) | Group 2: Unresectable Locally Advanced BCC (laBCC)
Number analyzed (Participants) | 54 | 84
mg/L
  Cycle 1 Day 1: number analyzed (Participants) | 47 | 81
  Cycle 1 Day 1 | 103 (25.2) | 104 (45.5)
  Cycle 3 Day 1 | 160 (52.7) | 192 (91.6)

15. Secondary Outcome: Number of Participants With Anti-Drug Antibody (ADA) Status
Description: Immunogenicity was characterized by ADA responses & titers. Responses categories: Negative - ADA negative response at all time points, regardless of missing samples; Pre-existing immunoreactivity - ADA positive response at baseline with all post first dose negative results or positive response at baseline with all post first dose ADA responses < 9-fold over baseline titer levels; Treatment-boosted response - positive response in the assay post first dose, ≥ 9-fold over baseline titer levels, when baseline results are positive; Treatment-emergent response - ADA positive response in the cemiplimab ADA assay post first dose when baseline results = negative or missing.
Time Frame: Cycle 1: Days 1 and 43; Cycles 3 and 5: Day 1 (Each cycle of 9 weeks)
Population: The anti-drug antibody set included all participants who received cemiplimab and who had at least 1 non-missing result in the ADA assay after the first dose of the study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Metastatic BCC (mBCC) | Group 2: Unresectable Locally Advanced BCC (laBCC)
Number analyzed (Participants) | 52 | 81
Participants
  Negative ADA | 50 | 74
  Pre-Existing ADA | 2 | 2
  Treatment-emergent ADA | 0 | 5

ADVERSE EVENTS:
Time Frame: From signature of informed consent until 105 days after last dose of study drug (up to 2129 days)
Arm/Group | Group 1: Metastatic BCC (mBCC) | Group 2: Unresectable Locally Advanced BCC (laBCC)
All-Cause Mortality (participants affected / at risk) | 22/54 | 21/84
Serious Adverse Events (participants affected / at risk) | 18/54 | 33/84
Other Adverse Events (participants affected / at risk) | 50/54 | 76/84
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: Metastatic BCC (mBCC) (N=54) | Group 2: Unresectable Locally Advanced BCC (laBCC) (N=84)
Urinary tract infection (Infections and infestations) | 1 (1) | 4 (4)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 1 (1) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 2 (3)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 2 (2) | 2 (2)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 2 (2)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1)
Autoimmune pericarditis (Cardiac disorders) | 1 (1) | 0 (0)
Autoimmune hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Immune-mediated hepatitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatitis C (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Oral candidiasis (Infections and infestations) | 0 (0) | 1 (1)
Soft tissue infection (Infections and infestations) | 0 (0) | 1 (1)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 1 (1)
Wound infection staphylococcal (Infections and infestations) | 0 (0) | 1 (1)
Arthritis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Atypical pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia staphylococcal (Infections and infestations) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Erosive oesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Brain oedema (Nervous system disorders) | 0 (0) | 1 (1)
Cerebrospinal fluid leakage (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 1 (2) | 1 (1)
Facial paralysis (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 2 (2)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 0 (0)
Autoimmune myocarditis (Cardiac disorders) | 1 (1) | 0 (0)
Immune-mediated myocarditis (Cardiac disorders) | 1 (1) | 0 (0)
Infected neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Brain neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lymphoproliferative disorder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Hypertensive crisis (Vascular disorders) | 0 (0) | 1 (2)
Peripheral ischaemia (Vascular disorders) | 0 (0) | 1 (1)
Phlebitis (Vascular disorders) | 0 (0) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 2 (2)
Hypophysitis (Endocrine disorders) | 0 (0) | 1 (1)
Lymphadenopathy mediastinal (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Dupuytren's contracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0)
Ear disorder (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (1)
General physical health deterioration (General disorders) | 1 (1) | 0 (0)
Sarcoidosis (Immune system disorders) | 0 (0) | 1 (2)
Radial head dislocation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Multiple fractures (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 1 (1)
Cachexia (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Delirium (Psychiatric disorders) | 0 (0) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Erysipelas (Infections and infestations) | 1 (1) | 0 (0)
Immune-mediated enterocolitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: Metastatic BCC (mBCC) (N=54) | Group 2: Unresectable Locally Advanced BCC (laBCC) (N=84)
Nausea (Gastrointestinal disorders) | 6 (9) | 13 (19)
Vomiting (Gastrointestinal disorders) | 7 (9) | 6 (10)
Constipation (Gastrointestinal disorders) | 12 (14) | 5 (6)
Diarrhoea (Gastrointestinal disorders) | 20 (26) | 20 (33)
Abdominal pain (Gastrointestinal disorders) | 4 (4) | 6 (7)
Anaemia (Blood and lymphatic system disorders) | 6 (7) | 13 (19)
Pyrexia (General disorders) | 7 (9) | 5 (7)
Asthenia (General disorders) | 5 (6) | 17 (27)
Fatigue (General disorders) | 24 (32) | 25 (35)
Oedema peripheral (General disorders) | 7 (9) | 5 (5)
Alanine aminotransferase increased (Investigations) | 3 (3) | 4 (6)
Blood creatinine increased (Investigations) | 4 (4) | 8 (9)
Decreased appetite (Metabolism and nutrition disorders) | 6 (6) | 14 (18)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (2) | 6 (12)
Hypokalaemia (Metabolism and nutrition disorders) | 4 (4) | 4 (6)
Hyperglycaemia (Metabolism and nutrition disorders) | 6 (8) | 2 (2)
Urinary tract infection (Infections and infestations) | 4 (5) | 10 (11)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 5 (6)
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 (10) | 16 (24)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 (9) | 4 (5)
Rash (Skin and subcutaneous tissue disorders) | 4 (4) | 6 (6)
Pruritus (Skin and subcutaneous tissue disorders) | 8 (13) | 20 (24)
Headache (Nervous system disorders) | 7 (8) | 12 (14)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 10 (14)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 11 (18)
Hypothyroidism (Endocrine disorders) | 4 (4) | 8 (9)
Influenza like illness (General disorders) | 2 (2) | 5 (7)
Pain (General disorders) | 3 (4) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 5 (6) | 7 (7)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 3 (3) | 7 (10)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 5 (6) | 6 (7)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 5 (6)
Eczema (Skin and subcutaneous tissue disorders) | 5 (7) | 5 (5)
Dry mouth (Gastrointestinal disorders) | 4 (4) | 3 (3)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 (3) | 5 (5)
Myalgia (Musculoskeletal and connective tissue disorders) | 5 (6) | 3 (3)
Neck pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 2 (4)
Bronchitis (Infections and infestations) | 0 (0) | 6 (7)
Upper respiratory tract infection (Infections and infestations) | 3 (3) | 6 (6)
Conjunctivitis (Infections and infestations) | 0 (0) | 5 (5)
Weight decreased (Investigations) | 5 (6) | 7 (7)
Blood creatine phosphokinase increased (Investigations) | 4 (5) | 6 (8)
Weight increased (Investigations) | 8 (12) | 2 (2)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 9 (12)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (5) | 8 (9)
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 5 (5)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 6 (6)
Dizziness (Nervous system disorders) | 5 (5) | 7 (8)
Hyperthyroidism (Endocrine disorders) | 5 (7) | 2 (2)
Hypertension (Vascular disorders) | 12 (33) | 9 (15)
Cataract (Eye disorders) | 0 (0) | 5 (6)
Fall (Injury, poisoning and procedural complications) | 4 (7) | 5 (5)
Infusion related reaction (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Anxiety (Psychiatric disorders) | 3 (3) | 3 (3)
Haematuria (Renal and urinary disorders) | 4 (5) | 3 (3)
Paraesthesia (Nervous system disorders) | 3 (3) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator has the right to independently publish study results from the investigator's site after a multi-center publication, or a defined period after the completion of the study by all sites. The investigator must provide the sponsor a copy of any such publication derived from the study for review and comment in advance of any submission, and delay publication, if requested, to allow the Sponsor to preserve its proprietary rights.

DOCUMENTS (2):
  • Study Protocol (2019-07-29): https://cdn.clinicaltrials.gov/large-docs/36/NCT03132636/Prot_000.pdf
  • Statistical Analysis Plan (2020-02-07): https://cdn.clinicaltrials.gov/large-docs/36/NCT03132636/SAP_001.pdf